CLINICAL TRIAL: NCT02244424
Title: Tools for Teen Moms: Reducing Infant Obesity Risk
Acronym: TFTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Mildred Horodynski, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21HDO75974-OIAL
Record Dates: First submitted 2014-06-24; First posted 2014-09-19 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Adolescent Mothers; Infant Obesity
Keywords: Infant; Obesity; Adolescent; Social media; Prevention
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tools for Teen Moms Intervention Group (Experimental): Tools for Teen Moms intervention group will receive daily challenges focusing on: 1) Maternal-Infant Feeding Interaction; and 2) Feeding Practices Challenges. The challenges will cycle through a pre-determined schedule where they are automatically updated each day at midnight. Participants will have a 24-hour period to complete each challenge. The intervention will provide a new daily challenge over six weeks, a time frame selected to provide participants with enough opportunities to form the habit of visiting the website daily. Participants will continue to receive usual MIHP care during the intervention.
  Interventions: Behavioral: Tools for Teen Moms
- MIHP standard care (No Intervention): MIHP care consists of voluntary home visits: one week postpartum, at six weeks, and six months, and on-going as needed provided by a RN, licensed social worker, RD, infant mental health specialist and/or paraprofessional. Content includes a flexible plan of care with visits based on identified domains for both the mother and the infant.

INTERVENTIONS:
Behavioral: Tools for Teen Moms — The Tools for Teen Moms intervention is a novel social media intervention platform designed by the investigators which includes cell phone text message reminders, and infant feeding website, and Facebook to increase infant-centered feeding through daily behavioral challenge activities ("challenges") for this population. The intervention consists of 6 weeks of daily challenges and will be delivered within the infant's first 6 months of life.
  Arms: Tools for Teen Moms Intervention Group

SUMMARY:
The purpose of this social media group randomized trial (GRT) is to test the feasibility of our Baby Dayr for Teen Moms intervention to increase maternal responsiveness to infant cues and implement healthy feeding practices through development of a healthy feeding style.

Aim 1: Evaluate the feasibility and acceptability of the Baby Dayr intervention administered to the target population as it relates to their acceptance and satisfaction with the content, format, delivery, and use of social media.

Aim 2: Explore efficacy of the Baby Dayr intervention administered to adolescent mothers of infants 4 months of age or less as assessed by maternal responsiveness, feeding style, and feeding practices evaluated at the completion of the intervention using self-report methods.

DETAILED DESCRIPTION:
Rapid weight gain during infancy is one of the strongest risk factors for obesity later in childhood. Weight gain in infancy is closely linked with feeding practices. Unhealthy mother-infant feeding practices contribute to rapid and/or excessive infant weight gain. Lower-income, adolescent, first-time mothers are less likely to engage in infant-centered feeding (ICF) which is characterized by maternal responsiveness (MR), healthy feeding styles (FS), and healthy feeding practices (FP). ICF is needed to reduce rapid/excessive weight gain during the first six months of life and to foster infant feeding self-regulation that is associated with healthy growth. ICF is a critical factor in reducing infant obesity risk and later adverse health conditions. Practical early intervention strategies are necessary to promote ICF among adolescent mothers to reduce obesity risk. We propose Baby Dayr, a novel social media intervention platform designed by the investigators which includes cell phone text message reminders, an infant feeding website, and Facebook to increase ICF through daily behavioral challenge activities ("challenges") for this population. Because cell phones permit natural, frequent and non-intrusive contact as they are not time-or-place-dependent, they offer an innovative strategy for intervening with adolescent mothers. However, this approach is untested for its feasibility with this population regarding infant feeding practices. We propose an exploratory, longitudinal, randomized, two-group study design. The three specific aims are: 1) to establish preliminary efficacy of the intervention as assessed by infant growth evaluated pre-intervention, immediately post intervention, and when the infant is six months old; 2) establish preliminary efficacy of the Baby Dayr plus Maternal-Infant Health Program (MIHP) care vs. MIHP care only on infant-centered feeding (MR, FS, and FP) mediated by maternal knowledge and self-efficacy; and 3) establish the feasibility, acceptability, and satisfaction of a social media intervention (Baby Dayr) for low-income adolescent, first-time mothers by assessing: 1) rates of enrollment and completion of daily challenges, 2) acceptability ratings of Baby Dayr; and 3) satisfaction with Baby Dayr. Participants will be randomly assigned to the intervention (Baby Dayr and MIHP) (n = 40) or control group (MIHP care only) (n = 40). The intervention consists of six weeks of daily challenges and will be delivered starting when the infant is four to six weeks old. The study is innovative in its: 1) assessment of ICF to reduce rapid/excessive infant weight gain in the first six months of life with low-income, adolescent, first-time mother-infant dyads, and 2) combination of an infant-centered skill-building, educational, and coaching approach using social media that is accessible and suitable for adolescents. The proposed research is significant in that it will contribute to the science related to ICF and knowledge regarding use of a social media platform in an at-risk population that can lead to reducing the risk of infant obesity. Information gained from this study will be used to refine the intervention for use in a larger-scale, longitudinal, randomized, controlled trial to reduce obesity risk in infants of low-income, adolescent mothers.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified, English-speaking
* Low-income, adolescent
* First-time mothers between the ages of 14 and 19
* With daily web access and access to a cell phone that includes text messaging capabilities
* Family income ≤ 185% of federal poverty
* Term birth (37≤42 weeks, 2500≤3750 grams birth weight)
* Mothers and infants with no special nutrients or feeding needs
* Infants less than six weeks old at study enrollment who have not started eating solid foods
* Adolescent mothers must be a primary caretaker of the infant who feeds her infant at least once a day, and who is willing to participate in a six-week intervention with data collection at three defined time points (T1, T2, and T3)

Exclusion Criteria:

* Male caregivers
* Mothers and infants with diagnosed feeding/eating disorders
* Significant perinatal or postnatal complications
* Post partum depression or other mental health problems
* Adolescent mothers who do not share in the feeding responsibility of their infants
* Adolescents without daily web access nor a cell phone with text messaging capabilities

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mildred A Horodynski, PhD, Principal Investigator — Michigan State University; Kami Silk, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Background] Horodynski MA, Silk K, Hsieh G, Hoffman A, Robson M. Tools for teen moms to reduce infant obesity: a randomized clinical trial. BMC Public Health. 2015 Jan 21;15:22. doi: 10.1186/s12889-015-1345-x. PMID 25604090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Teen mothers of infants were recruited. Teen mothers participated in the intervention. Infants were included for collection of demographic and weight data. Thus the actual number of participants is doubled to account for both the mothers and infants as participants. Protocol Enrollment number then is 164 ( 82 teen mothers and 82 infants).
Groups:
- Tools for Teen Moms Intervention Group: Tools for Teen Moms intervention group (N = 51 teen mothers) will receive daily challenges focusing on: 1) Maternal-Infant Feeding Interaction; and 2) Feeding Practices Challenges. The challenges will cycle through a pre-determined schedule where they are automatically updated each day at midnight. Participants will have a 24-hour period to complete each challenge. The intervention will provide a new daily challenge over six weeks, a time frame selected to provide participants with enough opportunities to form the habit of visiting the website daily. Participants will continue to receive usual MIHP care during the intervention.
  Tools for Teen Moms: The Tools for Teen Moms intervention is a novel social media intervention platform designed by the investigators which includes cell phone text message reminders, and infant feeding website, and Facebook to increase infant-centered feeding through daily behavioral challenge activities ("challenges") for this population.
- MIHP Standard Care: MIHP care consists of voluntary home visits: one week postpartum, at six weeks, and six months, and on-going as needed provided by a RN, licensed social worker, RD, infant mental health specialist and/or paraprofessional. Content includes a flexible plan of care with visits based on identified domains for both the mother and the infant. 31 teen mothers received MIHP standard care.
Period: Overall Study
Arm/Group | Tools for Teen Moms Intervention Group | MIHP Standard Care
Started (Teen mothers were the participants in the study; data were collected on their infants.) | 102 (Teens were the participants who received the intervention. Data were collected on the infants.) | 62 (Teen participants received the MIHP standard care. Data were collected on infants.)
Infants | 51 (Infants of participants included in the study for collection of demographic and weight data.) | 31 (Infants of participants included in the study for collection of demographic and weight data.)
Mothers | 51 | 31
Completed (Numbers include both mothers and infants in the study only.) | 82 (Data were collected on all of the infants of the teen moms (n = 41).) | 52 (Data were collected on all of the infants of teen moms (n = 26).)
Not Completed | 20 | 10
Not completed — Lost to Follow-up | 20 | 10

BASELINE CHARACTERISTICS:
Population: Both teen mothers and their infants were enrolled in the study. Teen mothers received the intervention and/or the standard care. Overall number of baseline participants is 164 (82 teen mothers and 82 infants). Data were collected for infants during the study. Baseline population demographics are provided for the teen mothers and infants.
Groups:
- Tools for Teen Moms Intervention Group: Tools for Teen Moms intervention group will receive daily challenges focusing on: 1) Maternal-Infant Feeding Interaction; and 2) Feeding Practices Challenges.
- Total: Total of all reporting groups
Arm/Group | Tools for Teen Moms Intervention Group | MIHP Standard Care | Total
Number analyzed (Participants) | 102 | 62 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  years
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 17.53 (1.30) | 17.61 (1.41) | 17.56 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Female | 51 | 31 | 82
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Hispanic or Latino | 18 | 14 | 32
    Not Hispanic or Latino | 33 | 17 | 50
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 22 | 12 | 34
    White | 24 | 17 | 41
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: teen mother participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  teen mother participants
    United States: number analyzed (Participants) | 51 | 31 | 82
    United States | 51 | 31 | 82
Marital Status [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Married | 4 | 3 | 7
    In a Relationship | 29 | 17 | 46
    Not in a Relationship | 18 | 11 | 29
Highest level of education completed [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    6th grade | 0 | 0 | 0
    7th grade | 2 | 1 | 3
    8th grade | 2 | 2 | 4
    9th grade | 2 | 2 | 4
    10th grade | 11 | 0 | 11
    11th grade | 16 | 13 | 29
    12th grade | 6 | 2 | 8
    High school diploma or GED | 11 | 7 | 18
    Completed some college credits | 1 | 3 | 4
    Missing | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Full time (at least 35 hours/week) | 3 | 0 | 3
    Working part-time | 3 | 4 | 7
    Not working | 45 | 27 | 72
Infant age at enrollment [Mean (Standard Deviation); unit: months] — Data on infant participants Population: Only infants were analyzed for this measure.
  months
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 1.21 (0.48) | 1.18 (0.54) | 1.20 (0.50)
Infant sex [Count of Participants; unit: Participants] — Data on infant participants Population: Only infants were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Male | 26 | 17 | 43
    Female | 25 | 14 | 39
Birth weight (kg) [Mean (Standard Deviation); unit: kg] — Data on infant participants Population: Only infants were analyzed for this measure.
  kg
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 3.21 (0.40) | 3.21 (0.43) | 3.21 (0.41)
Birth length (cm) [Mean (Standard Deviation); unit: cm] — Data on infant participants Population: Only infants were analyzed for this measure.
  cm
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 50.98 (2.71) | 50.70 (2.88) | 50.88 (2.77)
Infant Baseline weight (kg) [Mean (Standard Deviation); unit: kg] — Data on infant participants Population: Only infants were analyzed for this measure.
  kg
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 4.30 (0.75) | 4.27 (0.78) | 4.29 (0.76)
Infant Baseline length (cm) [Mean (Standard Deviation); unit: cm] — Data on infant participants Population: Only infants were analyzed for this measure.
  cm
    number analyzed (Participants) | 51 | 31 | 82
    (all) | 54.75 (2.99) | 55.05 (3.61) | 54.86 (3.22)
Breastfeeding status at baseline [Count of Participants; unit: Participants] — Data on teen mother participants Population: Only mothers were analyzed for this measure.
  Participants
    number analyzed (Participants) | 51 | 31 | 82
    Currently Breastfeeding | 18 | 16 | 34
    Breastfed in the past | 15 | 9 | 24
    Never Breastfed | 18 | 6 | 24
Solid feeding status at baseline [Count of Participants; unit: Participants] — Data on infant participants Population: This data pertains only to the infants.
  Participants
    Fed anything other than breastmilk or formula: number analyzed (Participants) | 51 | 31 | 82
    Fed anything other than breastmilk or formula: Yes | 0 | 1 | 1
    Fed anything other than breastmilk or formula: No | 51 | 30 | 81
    Fed anything other than breastmilk or formula: Missing | 0 | 0 | 0
    Given tastes of solid food from mother's finger: number analyzed (Participants) | 51 | 31 | 82
    Given tastes of solid food from mother's finger: Yes | 1 | 2 | 3
    Given tastes of solid food from mother's finger: No | 49 | 29 | 78
    Given tastes of solid food from mother's finger: Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Infant Growth
Description: Recumbent infant length (inches) and weight (pounds/ounces) measured at three separate time points. While recumbent infant length was collected in inches and weight collected in pounds/ounces, these measures were converted into z-score measurements for the outcome measurement of change in infant growth. Standardized weight scores are measures of relative weight adjusted for child age and sex. The z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A z-score of 0 is equal to the mean. Negative numbers indicated weight values lower than the mean and the positive numbers indicate weight values higher than the mean.
Time Frame: Baby is less than 2 months; baby is 3 months; baby is 6 months
Population: 82 participants were included in analysis at Time 1, 79 at Time 2, and 67 at Time 3. This is due to participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: Weight for age Z-score
Arm/Group | Tools for Teen Moms Intervention Group | MIHP Standard Care
Number analyzed (Participants) | 51 | 31
Weight for age Z-score
  Time 1 (infant 2-8 weeks of age) | -0.46 (0.90) | -0.44 (0.86)
  Time 2 (infant about 3 months): number analyzed (Participants) | 49 | 30
  Time 2 (infant about 3 months) | -0.33 (0.95) | -0.46 (0.93)
  Time 3 (infant about 6 months): number analyzed (Participants) | 41 | 26
  Time 3 (infant about 6 months) | -0.22 (1.17) | -0.21 (0.83)

ADVERSE EVENTS:
Arm/Group | Tools for Teen Moms Intervention Group | MIHP Standard Care
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/62
Other Adverse Events (participants affected / at risk) | 0/102 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No